CLINICAL TRIAL: NCT01126749
Title: An Open-Label, Multicenter, Randomized Phase Ib/II Study of Eribulin Mesylate Administered in Combination With Gemcitabine Plus Cisplatin Versus Gemcitabine Plus Cisplatin Alone as First-Line Therapy for Locally Advanced or Metastatic Bladder Cancer
Brief Title: Eribulin Mesylate Administered in Combination With Gemcitabine Plus Cisplatin Versus Gemcitabine Plus Cisplatin Alone as First-Line Therapy for Locally Advanced or Metastatic Bladder Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated as per sponsor's decision
Sponsor: Eisai Inc. (Industry)
Collaborators: PharmaBio Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-702; 2009-015915-42 (EudraCT Number)
Record Dates: First submitted 2010-05-17; First posted 2010-05-20 (Estimated); Results first posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-01

CONDITIONS: Bladder Cancer
Keywords: Locally Advanced or Metastatic Bladder Cancer, including other transitional cell cancers of the urothelium (prostate, urethra, ureter, and renal pelvis)
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; eribulin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E7389 in combination with gemcitabine plus cisplatin (Experimental)
  Interventions: Drug: Gemcitabine; Drug: E7389; Drug: Cisplatin
- gemcitabine plus cisplatin (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine
Drug: E7389 — E7389
  Other Names: Eribulin Mesylate
  Arms: E7389 in combination with gemcitabine plus cisplatin
Drug: Cisplatin — Cisplatin

SUMMARY:
The purpose of this study is to determine whether Patients with Locally Advanced or Metastatic Bladder Cancer who receive Eribulin Mesylate Administered in Combination with Gemcitabine Plus Cisplatin Versus Gemcitabine Plus Cisplatin Alone as First-Line Therapy is safety and tolerable when administered to patients with locally advanced or metastatic bladder cancer and to gain preliminary data on whether patients may benefit from this combination.

DETAILED DESCRIPTION:
This open-label, multicenter, randomized study will consist of 2 phases:

* Phase Ib: a safety run-in period with 3 ascending doses of eribulin;
* Phase II: a randomized 2-arm design. Phase Ib Patients will be recruited into cohorts, with a minimum of 3 and a maximum of 6 patients per cohort. All patients will receive the same dose of gemcitabine (1000 mg/m2 on Days 1 and 8 of a 21-day cycle) and cisplatin (70 mg/m2 on Day 1) in combination with eribulin (administered on Days 1 and 8 of the cycle). All patients in a cohort will receive the same dose level of eribulin.

The dose level of eribulin will be escalated for additional cohorts unless greater than 2 dose limiting toxicities (DLTs) are reported at the lower dose level(s) prior to enrollment of the next dose level. If one DLT occurs at any dose level, the cohort will be expanded to include up to a maximum of 6 patients.

A Dose Escalation Committee will determine when no further dose escalation is appropriate and whether the MTD will be defined as a preceding dose or an intermediate dose.

Phase II Patients will be randomized in a 1:1 ratio to receive either eribulin in combination with gemcitabine plus cisplatin (Arm 1) or gemcitabine plus cisplatin alone (Arm 2). The eribulin dose will be 1.0 mg/m2 administered on Days 1 and 8 of each 21-day treatment cycle, the recommended Phase II dose for eribulin when administered in combination gemcitabine plus cisplatin, as determined in the Phase Ib portion of the study.

Allocation of patients will be stratified based on metastatic disease status (patients with visceral metastases versus patients with non-visceral metastases). This stratified randomization will be centrally allocated across all centers via an Interactive Voice Activated Response System (IVRS).

For both the Phase Ib and Phase II portions, 1 cycle of therapy will last 21 days, with a maximum number of 6 gemcitabine plus cisplatin cycles. Radiologic examinations including a computed tomography (CT) scan of the chest, abdomen, and pelvis as appropriate (and CT or magnetic resonance imaging [MRI] scan as appropriate), will be performed during Screening and after every 6 weeks while on therapy. In the case of dose delays, scans should be performed according to the original Cycle 1 Day 1 schedule (ie, scans should not be delayed). Radiographic assessments should be repeated at withdrawal if the last assessment was obtained greater than 3 weeks from withdrawal of therapy. Patients will be followed until death following completion of therapy. Scans will be required every 2 months until documentation of PD or the start of a next line of therapy, whichever occurs first. In patients experiencing PD, follow-up will be for survival only and radiographic scans are not required.

ELIGIBILITY:
Inclusion Criteria

Patients may be entered in the study only if they meet all of the following criteria:

1. Male or female patient greater than 18 years of age;
2. Histologically or cytologically confirmed, locally advanced Stage 4 (eg, T4b) or metastatic transitional cell cancer of the bladder; including other transitional cell cancers of the urothelium (prostate, urethra, ureter, and renal pelvis)
3. Not previously treated with systemic chemotherapy for metastatic bladder cancer (one regimen of adjuvant or neoadjuvant chemotherapy is permitted). Patients must have a disease-free interval of 6 months after adjuvant therapy;
4. At least 1 site of measurable disease by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST version 1.1) guidelines;
5. Life expectancy of greater than or equal to 3 months;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1;
7. Patients must have active bowel function defined as at least 3 bowel movements per week according to subject history and must be willing to maintain a diary of bowel function prior to dosing and continuing through completion of study treatment. Laxatives may be used to maintain adequate bowel function;
8. Patients must have adequate renal function as evidenced by calculated creatinine clearance greater than or equal to 55 mL/min per the Cockcroft and Gault formula;
9. Patients must have adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L, hemoglobin greater than or equal to 10.0 g/dL (a hemoglobin less than 10.0 g/dL at Screening is acceptable if it is corrected to greater than or equal to 10.0 g/dL by growth factor or transfusion prior to first dose), and platelet count greater than or equal to 100 x 10^9/L;
10. Patients must have adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limit of the normal range (ULN), and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 x ULN (in the case of liver metastases, less than or equal to 5 x ULN). If there are bone metastases, liver-specific alkaline phosphatase may be separated from the total and used to assess liver function instead of total alkaline phosphatase;
11. Male or female patients of child-producing potential must agree to use double barrier contraception, oral contraceptives, or avoidance of pregnancy measures during the study and for 90 days after the last day of treatment;
12. Females of childbearing potential must have a negative serum pregnancy test at screening;
13. Females may not be breastfeeding;
14. Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria

Patients will not be entered in the study for any of the following reasons:

1. Prior treatment with epothilone, ixabepilone, patupilone, vinflunine, halichondrin B, and/or halichondrin B chemical derivatives;
2. History of other malignancies except: (1) adequately treated basal or squamous cell carcinoma of the skin; (2) curatively treated, a) in situ carcinoma of the uterine cervix, or b) prostate cancer, or c) superficial bladder cancer; or (3) other curatively treated solid tumor with no evidence of disease for greater than or equal to 3 years;
3. Presence of brain metastases, unless the patient has received adequate treatment at least 4 weeks prior to randomization, and is stable, asymptomatic, and off steroids for at least 4 weeks prior to randomization;
4. Received an investigational agent, chemotherapy, biological therapy, hormonal therapy, targeted therapy, or radiotherapy within 30 days prior to commencing study treatment, or have not recovered from all treatment-related toxicities to Common Toxicity Criteria (CTC) Grade less than or equal to 1, except for alopecia;
5. Are currently receiving an investigational agent or any other systemic anticancer treatment, including palliative radiotherapy;
6. Significant cardiovascular impairment (history of congestive heart failure New York Heart Association [NYHA] Grade greater than 2, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia);
7. Subjects with a high probability of Long QT Syndrome;
8. Patients with organ allografts requiring immunosuppression;
9. Known active infection with human immunodeficiency virus (HIV), hepatitis B, virus (HBV) or hepatitis C; virus (HCV);
10. Hypersensitivity to halichondrin B and/or halichondrin B chemical derivative
11. Prior pelvic radiation;
12. History of known or suspected peritoneal carcinomatosis with risk of bleeding or perforation, or intraluminal or serosal metastatic lesions with risk of bleeding or perforation of any lesions;
13. History of abdominal adhesions, fistula, diverticulitis, gastrointestinal perforation, intra-abdominal abscess, documented peptic ulcer disease (active gastroesophageal reflux disease/dyspepsia are allowed), or other gastrointestinal conditions with increased risk of perforation;
14. Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v.4.0) Grade greater than or equal to 2 constipation;
15. CTCAE v.4.0 Grade greater than or equal to 2 peripheral neuropathy;
16. Have any medical condition that would interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-04-16 (Actual); Primary Completion 2015-05-08 (Actual); Study Completion 2016-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (14):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Fort Myers, Florida
  - St. Petersburg, Florida
  - Ann Arbor, Michigan
  - Las Vegas, Nevada
  - East Orange, New Jersey
  - Rochester, New York
  - Chattanooga, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - Webster, Texas
  - Huntington, Virginia
  - Northfork, West Virginia
- Germany (7):
  - Aachen Northwest
  - Berlin
  - Essen, Northwest
  - Goch, Northwest
  - Hamburg, HH
  - Tuebingen, BW
  - Wiesbaden, HE
- Netherlands (3):
  - Maastricht
  - Nieuwegein
  - Nijmegen
- Spain (4):
  - Barcelona
  - Elche- Alicante
  - Madrid
  - Sabadell
- Ukraine (5):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lviv
- United Kingdom (5):
  - Leicester
  - Liverpool
  - London
  - Manchester
  - Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 32 investigative sites in Germany, Netherlands, Spain, Ukraine, United Kingdom and the United States from 16 April 2010 to 20 July 2016.
Pre-assignment Details: A total of 92 participants were enrolled in this study. This study consisted of two phases: Phase 1b and Phase 2. In Phase 1b, 9 participants were enrolled and received study treatment and in Phase 2, 83 participants were randomized, of which 80 participants received the study treatment.
Groups:
- Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2: Participants received Eribulin Mesylate 0.7 milligram per square meter (mg/m^2), as an intravenous infusion on Days 1 and 8 in combination with Gemcitabine 1000 mg/m^2, as an intravenous infusion on Days 1 and 8 and Cisplatin 70 mg/m^2, as an intravenous infusion on Day 1 of a 21-day cycle until the occurrence of disease progression (PD), unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, death, or for a maximum of six cycles of gemcitabine plus cisplatin (18 weeks), whichever occurred first.
- Phase 1b: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2: Participants received Eribulin Mesylate 1.0 mg/m^2, as an intravenous infusion on Days 1 and 8 in combination with Gemcitabine 1000 mg/m^2, as an intravenous infusion on Days 1 and 8 and Cisplatin 70 mg/m^2, as an intravenous infusion on Day 1 of a 21-day cycle until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, death, or for a maximum of six cycles of gemcitabine plus cisplatin (18 weeks), whichever occurred first.
- Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2: Participants received Eribulin Mesylate 1.0 mg/m^2 (Recommended Phase 2 dose), as an intravenous infusion on Days 1 and 8 in combination with Gemcitabine 1000 mg/m^2, as an intravenous infusion on Days 1 and 8 and Cisplatin 70 mg/m^2, as an intravenous infusion on Day 1 of each 21-day cycle until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, death, or for a maximum of six cycles of gemcitabine plus cisplatin (18 weeks), whichever occurred first.
- Phase 2: Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2: Participants received Gemcitabine 1000 mg/m^2, as an intravenous infusion on Days 1 and 8 and cisplatin 70 mg/m^2, as an intravenous infusion on Day 1 of each 21-day cycle until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, death, or for a maximum of six cycles of gemcitabine plus cisplatin (18 weeks), whichever occurred first.
Period: Phase 1b
Arm/Group | Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 1b: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2
Started | 3 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Death | 3 | 4 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 1b: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2
Started | 0 | 0 | 42 | 41
Safety Analysis Set (SAS)/Treated | 0 | 0 | 41 | 39
Modified-intent-to-treat (MITT) | 0 | 0 | 40 | 39
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 42 | 41
Not completed — Completed 1 Year Follow-Up Per Protocol | 0 | 0 | 4 | 7
Not completed — Study Termination by Sponsor | 0 | 0 | 12 | 6
Not completed — Other | 0 | 0 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 22 | 22
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: SAS included all participants who were randomized and treated in this study.
Groups:
- Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2: Participants received Eribulin Mesylate 0.7 mg/m^2, as an intravenous infusion on Days 1 and 8 in combination with Gemcitabine 1000 mg/m^2, as an intravenous infusion on Days 1 and 8 and Cisplatin 70 mg/m^2, as an intravenous infusion on Day 1 of a 21-day cycle until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, death, or for a maximum of six cycles of gemcitabine plus cisplatin (18 weeks), whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 1b: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Total
Number analyzed (Participants) | 3 | 6 | 41 | 39 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 15 | 14 | 35
  >=65 years | 1 | 2 | 26 | 25 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 5 | 7 | 14
  Male | 2 | 5 | 36 | 32 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 3 | 8
  Not Hispanic or Latino | 3 | 3 | 39 | 34 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 6 | 41 | 39 | 89
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicity (DLT) as Per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0
Description: DLTs were clinically significant adverse events within 21 days of treatment judged by investigator at least possibly related to treatment. This included greater than or equal to (>=) Grade 3 (G3) peripheral neuropathy, >=G3 nausea and vomiting despite optimal anti-emetic treatment, any other non-hematologic toxicity of >=G3 (except alopecia, single abnormal laboratory values the Investigator judged unlikely related to study therapy, had no clinical correlate, and resolved within 7 days, and hypersensitivity reaction to any of the compounds), Grade 4 neutropenia lasting over 7 days, febrile neutropenia (defined as fever >=38.5 degrees Celsius with absolute neutrophil count below 1.0*10^9 per liter, G3 thrombocytopenia with nontraumatic bleeding (without therapeutic systemic anticoagulation) requiring platelet transfusion, Grade 4 thrombocytopenia (with or without nontraumatic bleeding), any study drug-related death, any other toxicity the dose escalation committee believed to be DLT.
Time Frame: Cycle 1 (Cycle length=21 days)
Population: SAS included all participants who were randomized and treated in Phase 1b of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2 | Phase 1b: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2 + Cisplatin 70 mg/m^2
Number analyzed (Participants) | 3 | 6
Participants | 0 | 1

2. Primary Outcome: Phase 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE was defined as an adverse event that had an onset date, or a worsening in severity on or after the first dose of study drug up to the end of the study. Number of participants with TEAEs were reported based on safety assessments of laboratory tests, physical examination, examining bowel movements, regular measurement of vital signs, eastern cooperative oncology group-performance status and electrocardiogram parameter values. SAE was any untoward medical occurrence that at any dose: resulted in death; life threatening required inpatient hospitalization; resulted in persistent, significant disability; was congenital anomaly/birth defect or medically important due to other reasons than mentioned criteria. Number of participants with TEAEs and SAEs were reported.
Time Frame: From the first dose of study drug up to approximately 6 years 3 months
Population: SAS included all participants who were randomized and treated in Phase 2 of this study.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2: Participants received Eribulin Mesylate 1.0 mg/m^2 (Recommended Phase 2 dose), as an intravenous infusion on Days 1 and 8 in combination with Gemcitabine 1000 mg/m^2, as an intravenous infusion on Days 1 and 8 and Cisplatin 70 mg/m^2, as an intravenous infusion on Day 1 of each 21-day cycle until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, death, or for a maximum of six cycles of gemcitabine plus cisplatin (18 weeks), whichever occurred first.
- Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2: Participants received Gemcitabine 1000 mg/m^2, as an intravenous infusion on Days 1 and 8 and cisplatin 70 mg/m^2, as an intravenous infusion on Day 1 of each 21-day cycle until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, death, or for a maximum of six cycles of gemcitabine plus cisplatin (18 weeks), whichever occurred first.
Arm/Group | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2
Number analyzed (Participants) | 41 | 39
Participants
  TEAEs | 41 | 38
  SAEs | 22 | 14

3. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization until the earlier of the following two events: the date of disease progression (PD) or the date of death based on response evaluation criteria in solid tumor (RECIST) version (v) 1.1. PD was defined as at least a 20 percent (%) increase or 5 millimeter (mm) increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization until the earlier of the following two events: the date of PD or the date of death (Up to approximately 6 years 3 months)
Population: Modified intent-to-treat (MITT) analysis set included all participants who were randomized and received at least one dose of study medication without major protocol eligibility violations. Due to the lack of a clear definition for PFS censoring rules and deviation from the statistical analysis plan relating to interim analyses, the PFS analysis was deemed unreliable and therefore data was not collected and reported.
Arm/Group | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 2: Percentage of Participants With Overall Response
Description: Overall response rate was defined as the percentage of participants with the best confirmed response of complete response (CR) or partial response (PR) based on RECIST v1.1. CR was defined as complete disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline summed longest diameters.
Time Frame: From the date of randomization until CR or PR (Up to approximately 6 years 3 months)
Population: MITT analysis set included all participants who were randomized and received at least one dose of study medication without major protocol eligibility violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2
Number analyzed (Participants) | 40 | 39
percentage of participants | 52.5 [37.0 to 68.0] | 46.2 [30.5 to 61.8]

5. Secondary Outcome: Phase 2: Percentage of Participants With Progression-free Survival at Week 12
Description: PFS was defined as the time from the date of randomization until the earlier of the following two events: the date of PD or the date of death based on RECIST v1.1. PD was defined as at least a 20% increase or 5 mm increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: Week 12
Population: MITT analysis set included all participants who were randomized and received at least one dose of study medication without major protocol eligibility violations. Due to the lack of a clear definition for PFS censoring rules and deviation from the statistical analysis plan relating to interim analyses, the PFS analysis was deemed unreliable and therefore data was not collected and reported.
Arm/Group | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: TTP was defined as the time from the date of randomization until the date of PD based on RECIST v1.1. PD was defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking in reference the smallest summed longest diameters on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of 1 or more new lesions was also considered progression.
Time Frame: From the date of randomization until the date of PD (Up to approximately 6 years 3 months)
Population: as for outcome 5
Arm/Group | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death due to any cause.
Time Frame: From the date of randomization until the date of death (Up to approximately 6 years 3 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2
Number analyzed (Participants) | 40 | 39
weeks | 62.9 [39.86 to 132.0] | 64.6 [50.43 to 126.4]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to approximately 6 years 3 months
Description: SAS included all participants who were randomized and treated in this study.
Groups:
- Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2: Participants received Eribulin Mesylate 0.7 mg/m^2, as an intravenous infusion on Days 1 and 8 in combination with Gemcitabine 1000 mg/m^2, as an intravenous infusion on Days 1 and 8 and Cisplatin 70 mg/m^2, as an intravenous infusion on Day 1 of a 21-day cycle until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, death, or for a maximum of six cycles of gemcitabine plus cisplatin (18 weeks), whichever occurred first.
- Phase 1b: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2: Participants received Eribulin Mesylate 1.0 mg/m^2, as an intravenous infusion on Days 1 and 8 in combination with Gemcitabine 1000 mg/m^2, as an intravenous infusion on Days 1 and 8 and Cisplatin 70 mg/m^2, as an intravenous infusion on Day 1 of a 21-day cycle until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, death, or for a maximum of six cycles of gemcitabine plus cisplatin (18 weeks), whichever occurred first.
Arm/Group | Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 | Phase 1b: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 | Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/6 | 22/41 | 22/39
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 22/41 | 14/39
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 41/41 | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 (N=3) | Phase 1b: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 (N=6) | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 (N=41) | Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Small Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 5 (7)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant Nipple Neoplasm Male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Eribulin Mesylate 0.7 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 (N=3) | Phase 1b: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 (N=6) | Phase 2: Eribulin Mesylate 1.0 mg/m^2 + Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 (N=41) | Phase 2: Gemcitabine 1000 mg/m^2+ Cisplatin 70 mg/m^2 (N=39)
Anaemia (Blood and lymphatic system disorders) | 3 (7) | 5 (14) | 22 (30) | 22 (34)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 12 (41) | 7 (22)
Neutropenia (Blood and lymphatic system disorders) | 3 (13) | 3 (21) | 25 (82) | 19 (60)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (10) | 5 (22) | 18 (41) | 14 (36)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (5) | 5 (5) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (7) | 4 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 2 (4) | 15 (21) | 15 (16)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 12 (23) | 12 (20)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (7) | 6 (13) | 26 (45) | 26 (52)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 9 (14) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (9) | 12 (23) | 19 (30)
Asthenia (General disorders) | 2 (2) | 2 (8) | 12 (32) | 13 (29)
Chills (General disorders) | 0 (0) | 2 (5) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (7) | 5 (19) | 19 (30) | 20 (33)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (3) | 1 (1) | 4 (4) | 3 (4)
Pyrexia (General disorders) | 2 (5) | 2 (3) | 9 (17) | 6 (6)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 3 (4)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2) | 6 (7) | 5 (7)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (9) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (10) | 6 (37) | 10 (39)
Platelet count decreased (Investigations) | 0 (0) | 1 (4) | 7 (18) | 8 (16)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 3 (3) | 5 (6)
White blood cell count decreased (Investigations) | 0 (0) | 1 (11) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 5 (12) | 12 (20) | 21 (26)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 7 (8) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 3 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6) | 7 (7) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 3 (3) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 4 (6) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 4 (4) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0) | 5 (7) | 5 (5)
Dysaesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 11 (12) | 9 (13)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 4 (5) | 3 (4)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 4 (7) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 5 (8) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) | 6 (9)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (3) | 5 (5)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 4 (4) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 16 (17) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 4 (5)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ototoxicity (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 4 (5)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood magnesium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 3 (6) | 1 (2)
Endoscopy upper gastrointestinal tract abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (7) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (7)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphatic system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (6)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital lesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Social problem (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasodilatation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the lack of a clear definition for PFS censoring rules and deviation from the statistical analysis plan relating to interim analyses, the PFS analysis was deemed unreliable and therefore data was not collected and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes